CLINICAL TRIAL: NCT05871905
Title: [14 C] Study on Mass Balance of TY-9591 in Healthy Chinese Adult Male Subjects
Brief Title: [14 C] Study on Mass Balance of TY-9591 in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1601103
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TY-9591 (Experimental): TY-9591
  Interventions: Drug: TY-9591

INTERVENTIONS:
Drug: TY-9591 — C14 TY-9591
  Other Names: C14 TY-9591

SUMMARY:
[14 C] Mass balance clinical trial of TY-9591 in healthy Chinese subjects

DETAILED DESCRIPTION:
This is a single-center, non-randomized, one-arm, open trial in healthy adult subjects. The study population is male healthy subjects. The trial consisted of a screening period, a trial period and a follow-up period. A total of 6-10 healthy Chinese adult male subjects were planned to be enrolled and divided into groups according to specific conditions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be at least 50.0 kg in weight, and have a body mass index (BMI) in the range of 18.0-30.0 [BM= weight (kg)/ height 2(m)] (including the critical value.

  2.Subjects were sterile themselves, or voluntarily took highly effective non-drug contraception or abstained from sex completely from the beginning of self-medication to 1 year after administration.

  3.Volunteer to participate and sign informed consent, be able to communicate well with the investigator and complete the investigator in accordance with the study regulations.

Exclusion Criteria:

* 1.After a thorough physical examination, vital signs, routine laboratory tests (blood routine, blood biochemistry, coagulation function). Urine routine, stool routine + occult blood), anal digital examination, thyroid function, 12-lead electrocardiogram, chest X-ray (positive position), abdominal color Doppler ultrasound, liver, bile, pancreas, spleen and kidney) and other tests with clinical significance.

  2.Abnormal ophthalmic examination (intraocular pressure, slit lamp, fundus film) with clinical significance.

  3.Test positive for either hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antigen/antibody, or syphilis antibo.

  4.Those who smoked more than 5 cigarettes a day or habitually used nicotine products in the 3 months before screening, or were unable to abstain during the trial.

  5.A history of severe diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal system, respiratory system, metabolism and bone system, or any other disease or physiological condition that may affect the results of the study.

  6.Who participated in any drug clinical trial as a subject within 3 months prior to the administration of this trial.

  7.Those who had taken any prescription, over-the-counter, herbal and health products in the 14 days prior to screening.

  8.Those who cannot tolerate venous puncture blood collection or fainting blood or fainting needle.

  9.Those who have special dietary requirements and fail to follow the diets and regulations provided.

  10.The investigator considers it inappropriate to participate in clinical trials or is otherwise unable to complete the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
The total radioactivity in whole blood and plasma after a single oral administration of 14C TY-9591 | After oral administration of 14C TY-9591, the radiometabolite profiles of plasma, urine and stool were obtained to identify the major metabolites
  The total radioactivity in excreta after oral administration of 14C TY-9591

SECONDARY OUTCOMES:
The concentrations of TY-9591 by the verified LC-MS/MS method to obtain the pharmacokinetic parameters of TY-9591 and its metabolites D1 and D2 or ot | 8m
  To observe the safety of 14C TY-9591 in healthy subjects after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Mu Liyan, Principal Investigator — Suzhou First People's Hospital
Locations (1):
- Suzhou first people's hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No